CLINICAL TRIAL: NCT03945474
Title: Osteopathic Manipulative Treatment(OMT) for the Management of Feeding Dysfunction in Breastfed Newborns
Brief Title: Osteopathic Manipulation in Breastfed Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Methodist Medical Center of Illinois (Other)
Collaborators: University of Illinois College of Medicine at Peoria (Other); OSF Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 986099
Record Dates: First submitted 2019-04-23; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Osteopathic Medicine; Breast Feeding
MeSH Terms: conditions — Breast Feeding | interventions — salicylhydroxamic acid; Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either arm, OMT or sham.
Who Masked: Participant, Care Provider
Masking Description: Parents, infants and lactation consultants are not made aware of in which group the patient is placed, OMT or sham. Physicians are the only people aware of treatment/sham status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT (Experimental): Patients will receive a standardized protocol of: condylar decompression, Still's technique for the sternocleidomastoid, hyoid rebalancing and thoracic inlet myofascial release.
  Interventions: Other: Osteopathic Manipulation, OMT
- Sham (Sham Comparator): Patient will be treated in the supine position, with hands gently applied without pressure to the four areas: occiput, lateral cervical spine, hyoid area and thoracic inlet.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Sham — See description in sham arm.
  Arms: Sham
Other: Osteopathic Manipulation, OMT — See description in OMT arm
  Arms: OMT

SUMMARY:
Osteopathic manipulative treatment(OMT) is a form of manual medicine in which a trained physician uses his or her hands to diagnose areas of restriction in a patient's body. The physician then uses his or her hands to manually correct the restriction, to improve body function. The research team will be performing OMT on breastfed newborns that have been identified by lactation consultants as having a feeding issues. The team will then compare the feeding behaviors of these babies to those in the same category who did not receive OMT. OMT has some similarities to chiropractic manipulation. No thrusting techniques that produce a popping or cracking sound, as traditionally associated with chiropractic, will be used in this study.

Infants will be assigned to either the OMT group or No OMT group by the research team using a randomized process to help ensure equal enrollment in both groups. All babies will receive standard lactation support. All newborns receiving OMT will undergo the same four treatments, all of which involve light touch and massage. All newborns not receiving OMT will undergo a gentle application of light touch but no treatment. OMT treatment or sham sessions will be brief, taking no longer than 10 minutes, with each infant receiving two sessions during the study. During breastfeeding sessions, a lactation consultant will assess the infant's breastfeeding behavior using a tool called the LATCH score. He/she will be scored upon enrolling in the study, daily during hospitalization and before discharge from the hospital. The breastfeeding scores of the newborns who received OMT will be compared to the scores of those who did not.

The following is information regarding the types of treatment the investigators will use in the study:All treatments will be done with the baby lying on his or her back and will be gentle, applying no more force than would be used to test a tomato for ripeness. The provider's touch will be delicate enough so as not to blanch his or her fingernail beds while treating the infant. The first technique will reduce tightness in the sternocleidomastoid muscle, a front neck muscle that bends the head to one side and rotates the head the opposite side. The second technique treatment is used to correct tightness at the occipital condyle, which is the joint formed by the bone at the base of the skull and the top vertebrae of the neck. The hyoid bone is located in the neck and it aids in tongue movement and swallowing. The practitioner will apply gentle motion to the hyoid bone, usually using a finger and thumb. In the last technique, the physician will apply gentle motion to the connective tissue circling the baby's upper chest, shoulders, upper back, and lower neck, typically using the thumb and a few fingers on each hand. The purpose of this study is to determine whether osteopathic manipulative treatment (OMT) as an adjunct to lactation support will improve outcomes in breastfed newborns with feeding dysfunction.

DETAILED DESCRIPTION:
This project is an IRB-approved, single-blinded, randomized, controlled, prospective study that is currently taking place at two hospitals in Central Illinois. Inclusion criteria includes: term infants > 37 weeks gestation in the Level I nursery receiving lactation support and identified by lactation as having a newborn component to feeding dysfunction, who must be available for at least two inpatient treatment sessions and whose parent has provided informed consent.

All breastfed mother-infant dyads are offered evaluation by a lactation consultant. Breastfeeding sessions are routinely scored by either registered nurses or lactation consultants using the LATCH tool, with scores entered into a flowsheet on the electronic medical record. LATCH is a validated tool designed by Jensen et al to evaluate five components of breastfeeding: latch, audible swallowing, type of nipple, comfort of mother, and help mother needs holding infant to breast. For the purposes of the study, the nipple component will be excluded, so the maximum score will be 8. Eligible infants are enrolled in the study by a lactation consultant, who then notifies an on-call physician. The infant's mother is provided with a brochure explaining OMT and outlining potential benefits in newborns. The on-call physician provides informed consent and performs either the OMT or sham protocol. Infants are enrolled Monday through Thursday, and treatments are performed Monday through Friday. Enrolled infants are added to a password-protected, numerical list and randomized into their group based upon whether they land on an even number (sham) or an odd number (OMT). If multiple infants are enrolled at the same time, they are added to the list in alphabetical order. Group assignments are blinded to the parents, nursing staff, and lactation consultants. A brief note acknowledging that the infant has been enrolled in the study is entered into the electronic medical record. The OMT/sham treatments are documented on paper; kept in a locked document folder in the residency teaching clinic; and scanned into the electronic medical record two weeks after discharge.

The OMT treatment protocol includes the following four techniques: condylar decompression, cervical Still technique, thoracic inlet release and balancing of the hyoid bone. Infants in the control arm receive "sham" OMT during which they receive a gentle application of light touch but no treatment. A research team physician follows up on the day following enrollment to provide a second treatment. After discharge, each enrolled infant's LATCH scores are reviewed and documented.

Based upon results of smaller studies, the investigators hypothesize that infants receiving OMT in the treatment arm of the study will have more significant improvement in their LATCH score compared to infants in the control arm of the study receiving lactation support alone.

ELIGIBILITY:
Inclusion Criteria:

* term infants > 37 weeks gestation
* Level I newborn
* receiving lactation support
* identified by lactation as having a newborn component to feeding dysfunction, -must be available for at least two inpatient treatment sessions
* parent has provided informed assent.

Exclusion Criteria:

* infants <37 weeks gestation
* Level II or III nursery status
* wards of the state
* receiving speech or physical therapy
* currently receiving OMT, bottlefed infants
* infants breastfeeding with maternal factors contributing to feeding dysfunction (e.g. nipple problem).

Ages: 20 Hours to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Latch Score | Every feeding from birth until first treatment, up to 3 days of life
  LATCH is a 10 point scale that attaches 2 points to 5 measures: L(latch): 0=too sleep, no latch, 1=repeated attempts, hold nipple in mouth, 2=grasps breast, tongue down, lips placement and sucking pattern. A(audible swallowing): 0=none, 1=a few with stimulation, 2=spontaneous and intermittent. T(type of nipple): excluded due to maternal factors. C(comfort of breast/nipple):0=engorged, cracked, bleeding, severe discomfort, 1=filling small blisters, mild-mod discomfort, 2= soft, tender. H(hold of infant): 0=full assist by staff, 1=minimal assist, teach one side and mother does other side, 2=no assistance, Mother positions and holds infant swallowing, comfort, hold. This study uses a subscale without the T(nipple type). The total range of the LATCH scores will be 0-8, with 8 being the highest score, indicating successful breastfeeding. A score of 0 indicates poor breastfeeding.
Latch Score | from OMT/Sham until discharge or followup with lactation(4 weeks of life)
  LATCH is a 10 point scale that attaches 2 points to 5 measures: L(latch): 0=too sleep, no latch, 1=repeated attempts, hold nipple in mouth, 2=grasps breast, tongue down, lips placement and sucking pattern. A(audible swallowing): 0=none, 1=a few with stimulation, 2=spontaneous and intermittent. T(type of nipple): excluded due to maternal factors. C(comfort of breast/nipple):0=engorged, cracked, bleeding, severe discomfort, 1=filling small blisters, mild-mod discomfort, 2= soft, tender. H(hold of infant): 0=full assist by staff, 1=minimal assist, teach one side and mother does other side, 2=no assistance, Mother positions and holds infant swallowing, comfort, hold. This study uses a subscale without the T(nipple type). The total range of the LATCH scores will be 0-8, with 8 being the highest score, indicating successful breastfeeding. A score of 0 indicates poor breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique K Fons, MD, Principal Investigator — Methodist Medical Center of Illinois
Locations (2):
- United States (2):
  - UnityPoint Methodist Peoria Medical Center, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pizzolorusso G, Cerritelli F, D'Orazio M, Cozzolino V, Turi P, Renzetti C, Barlafante G, D'Incecco C. Osteopathic evaluation of somatic dysfunction and craniosacral strain pattern among preterm and term newborns. J Am Osteopath Assoc. 2013 Jun;113(6):462-7. PMID 23739757
- [Background] Pizzolorusso G, Turi P, Barlafante G, Cerritelli F, Renzetti C, Cozzolino V, D'Orazio M, Fusilli P, Carinci F, D'Incecco C. Effect of osteopathic manipulative treatment on gastrointestinal function and length of stay of preterm infants: an exploratory study. Chiropr Man Therap. 2011 Jun 28;19(1):15. doi: 10.1186/2045-709X-19-15. PMID 21711535
- [Background] Riordan J, Bibb D, Miller M, Rawlins T. Predicting breastfeeding duration using the LATCH breastfeeding assessment tool. J Hum Lact. 2001 Feb;17(1):20-3. doi: 10.1177/089033440101700105. PMID 11847847
- [Background] Herzhaft-Le Roy J, Xhignesse M, Gaboury I. Efficacy of an Osteopathic Treatment Coupled With Lactation Consultations for Infants' Biomechanical Sucking Difficulties. J Hum Lact. 2017 Feb;33(1):165-172. doi: 10.1177/0890334416679620. Epub 2016 Dec 27. PMID 28027445
- [Background] Kumar SP, Mooney R, Wieser LJ, Havstad S. The LATCH scoring system and prediction of breastfeeding duration. J Hum Lact. 2006 Nov;22(4):391-7. doi: 10.1177/0890334406293161. PMID 17062784
- [Background] Lund GC, Edwards G, Medlin B, Keller D, Beck B, Carreiro JE. Osteopathic manipulative treatment for the treatment of hospitalized premature infants with nipple feeding dysfunction. J Am Osteopath Assoc. 2011 Jan;111(1):44-8. doi: 10.7556/jaoa.2011.111.1.44. PMID 21258016
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525

DOCUMENTS (2):
  • Informed Consent Form (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT03945474/ICF_000.pdf
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT03945474/Prot_001.pdf